CLINICAL TRIAL: NCT04182646
Title: A Clinical Study on the Effect of Adjustable Intragastric Balloon in Obese Patients With Non Alcoholic Fatty Liver Disease(NAFLD) or Non-Alcoholic Steatohepatitis (NASH) With or Without Diabetes Mellitus
Brief Title: Effect of Adjustable Intragastric Balloon in Obese Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Rakesh Kalapala, Consultant Gastroenterologist, Asian Institute of Gastroenterology, India
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIG-G/IGBFLP
Record Dates: First submitted 2019-08-03; First posted 2019-12-02 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2021-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non-Alcoholic Steatohepatitis; Obesity; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The Spatz Adjustable intragastric balloon (AIGB) was developed to extend implantation to 1 year which have capability for decrease balloon volume for intolerance and increase volume for diminishing weight loss effect. The concept of an adjustable balloon came from the fact that around 10% of patients are intolerant to the balloon, requiring early extraction and also gastric balloons lose their effectiveness by approximately the 4th month post-implantation, and studies have shown that patients actually regain weight while the balloon is still implanted. AIGB balloon can mitigate this effect by adjustment of balloon volumes as required
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): The Spatz Adjustable intragastric balloon (AIGB) was developed to extend implantation to 1 year, decrease balloon volume for intolerance and increase volume for diminishing weight loss effect. The concept of an adjustable balloon came from the fact that around 10% of patients are intolerant to the balloon, requiring early extraction and also gastric balloons lose their effectiveness by approximately the 4th month post-implantation, and studies have shown that patients actually regain weight while the balloon is still implanted. AIGB balloon can mitigate this effect by adjustment of balloon volumes as required.
  Interventions: Device: Spartz Balloon

INTERVENTIONS:
Device: Spartz Balloon — The Spatz Adjustable intragastric balloon (AIGB) was developed to extend implantation to 1 year, decrease balloon volume for intolerance and increase volume for diminishing weight loss effect. The concept of an adjustable balloon came from the fact that around 10% of patients are intolerant to the balloon, requiring early extraction and also gastric balloons lose their effectiveness by approximately the 4th month post-implantation, and studies have shown that patients actually regain weight while the balloon is still implanted. AIGB balloon can mitigate this effect by adjustment of balloon volumes as required

SUMMARY:
Aims and objectives:

The Investigator aimed to evaluate effect of adjustable intra gastric balloon on non-alcoholic fatty liver disease/non alcoholic steatohepatitis (NAFLD/NASH) with or without diabetes mellitus, who have failed to achieve >10% of total body weight with lifestyle interventions and pharmacotherapy for weight loss.

The Investigator will evaluate NASH parameters such as NASH activity score(NAS), liver function tests along with weight loss and change in glycaemic control and changes in hormonal activity.

Sample size:

Based on previous study, to achieve median reduction of 40% in NAS score with 80% power and 0.05 as type 1 error; total sample size required is 36 cases.

DETAILED DESCRIPTION:
Introduction:

Nonalcoholic fatty liver disease (NAFLD) is an emerging major health problem worldwide which affects a significant proportion of the western population and there is gradual spread of this epidemic to south-east Asian countries. NAFLD encompasses two entities: Non-alcoholic fatty liver (NAFL) and Non-alcoholic steatohepatitis (NASH). NAFL is defined as the evidence of hepatic steatosis without inflammation either by raised liver enzymes, imaging or by histology in individuals without significant alcohol consumption in whom secondary causes of steatosis are absent. NASH on the other hand, is characterized by the presence of both steatosis and inflammation with evidence of hepatocyte injury in the form of ballooning with or without fibrosis.

Materials and Methods:

Study Enrollment:

Participants with diabetes attending the liver and bariatric clinic of the institute who have a Body Mass Index (BMI) > 27.5 Kg/m2 would be screened for eligibility. At first diagnosis of NAFLD / NASH, participants would be advised as per protocol to first attend the department of dietetic and nutrition for a low calorie diet and would also be advised for life style modifications for the next 6 months. They would be explained that the target weight loss would be 10% of the base weight. The exercise program would include a combination of aerobic, resistive and core building exercises. The participants would also be screened for secondary causes of obesity like hypothyroidism, hypercortisolism etc. Co morbidities like hypertension, hypothyroidism etc. would be screened and treated accordingly as per protocol. Secondary causes of NAFLD/ NASH would be ruled out by adequate history of intake of any steatogenic drugs as well as ruling out other conditions like Wilson disease, Autoimmune hepatitis, Viral hepatitis etc. Baseline investigations would include complete hemogram , liver function tests, anti-nuclear antibodies, anti-smooth muscle antibodies, anti-liver-kidney-microsomal antibodies, serum copper, serum ceruloplasmin, thyroid stimulating hormone , 8 am serum cortisol, fasting insulin, hepatitis B surface antigen and anti-hepatitis C antibody screening. Additional tests would include renal function tests, gut hormones assessment, electrocardiography, ultrasonography of the abdomen with acoustic resonance fibrosis imaging (ARFI) or a fibro scan. Additional tests like CT abdomen or high density proton fraction estimation by Magnetic resonance imaging would be done wherever clinically indicated. A liver biopsy would be advised to assess the presence of NASH and grading of fibrosis would be done by the interventional radiologist and reported by expert pathologist.

Follow-up:

At the 3rd month visit, participants would be re motivated and re-explained the weight loss importance and the lifestyle and dietary changes for resolution of NAFLD/ NASH. At this stage, they would be introduced the concept of endoscopic intragastric balloon as a prospective treatment as a part of the clinical study.

At the 6-month visit, if the participants has failed to lose at least 7% weight despite adequate exercise and lifestyle and dietary changes, then they would be offered to be enrolled in this clinical study. Alternative therapies including bariatric surgery and continuing with life style modifications and medications would be explained.

Method of Balloon Insertion and Post Procedure Care:

All participants will undergo upper gastrointestinal endoscopy using conscious sedation with or without an anaesthetist using one or more of the following medications - Propofol or midazolam.

The Spatz balloons are usually inflated with a mean 450ml (400-500ml) of normal saline with the addition of 2-3 ml of a 1% solution of Methylene Blue. After the 5th post-procedure day, a progressive full liquid to soft solid 1,200-1,400 kcal diet will be started. At one month follow up with principal investigator will be done. Participants who are intolerant to the balloon could be adjusted downward by 50-100 ml. Participants with one or more of the following were offered upward adjustments of the balloon volume (100-200 ml at the discretion of the endoscopist): weight loss plateau; lack of balloon effect; ability to overeat without resultant symptoms (any of the following: nausea, vomiting, bloating, eructation, abdominal pain, acid reflux symptoms). After 12 months of placement, the balloon will be deflated by aspiration via catheter and then retrieved under endoscopic/fluoroscopic guidance.

The data will be collected in excel sheets and later analysed using statistical analysis software. Any adverse effects would be noted and any serious adverse effects like severe pain, severe diarrhoea or catheter impaction which has been reported in less than 1% participants would be reported and adequate measures will be taken.

ELIGIBILITY:
Inclusion Criteria:

1. Participants (age 18- 65) diagnosed to have NAFLD / NASH as per imaging and histological criteria of American Association for Study of Liver Diseases (AASLD) with or without Diabetes Mellitus and who have failed the non-invasive approach to weight loss within the last 6 months. This would include patients who have failed to lose at least 10% of their base weight with dietary and lifestyle changes along with pharmacotherapy.
2. Patients with BMI > 27.5 kg/m2 who are unable to tolerate exercise program for weight loss.
3. Patients with BMI > 32.5 Kg/m2 who have NAFLD / NASH but are not willing for bariatric surgery.

Exclusion Criteria:

1. Previous history of gastric or bariatric surgery
2. Current or recent (within 6 months) gastric or duodenal ulcers
3. Cirrhosis patients with clinically significant portal hypertension defined as Hepatic Venous Pressure Gradient (HVPG) > 12 or recent variceal or Portal hypertensive gastropathy related bleed within the last 3 months
4. Presence of inflammatory disease of the gastrointestinal tract including esophagitis, gastric ulceration, duodenal ulceration, cancer or specific inflammation such as Crohn's disease.
5. A large hiatal hernia or >5 cm hernia or ≤5 cm with associated severe or intractable gastro-esophageal reflux symptoms.
6. Achalasia or any other severe motility disorder that may pose a safety risk during removal of the device.
7. Any gastric space occupying lesions including polyps,
8. Patients who are known to have or suspected to have an allergic reaction to materials contained in Adjustable balloon.
9. Psychologically unstable patients or patients with known psychiatric illness.
10. Patients unwilling to participate in an established medically-supervised diet and behaviour modification program, with routine medical follow-up.
11. Patients receiving aspirin, anti-inflammatory agents, anticoagulants or other gastric irritants, not under medical supervision.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Change in NAFLD activity Score | 6 months
  The 'NAFLD activity score' (NAS) is the most widely used histological grading and staging system for NAFLD. It is a histological scoring system addressing the full spectrum of NAFLD. It includes steatosis, hepatocellular ballooning, lobular inflammation, fibrosis, and the absence of lipogranulomas. In our study, liver histology was assessed by a single pathologist before and after treatment.
  Steatosis is graded as 0, 1, 2 and 3 depending on steatosis in hepatocytes.Lobular inflammation is graded as 0,1,2 and 3 depending on number of foci of inflammation per 20x field. Hepatocellular ballooning is graded as 0,1 and 2 depending on amount of ballooning. Fibrosis is graded as 0,1,2,3 and 4 depending on level of fibrosis. A composite score is calculated by addition on individual scores from steatosis, hepatocellular ballooning, lobular inflammation and fibrosis.

SECONDARY OUTCOMES:
Mean Percentage of Total Body Weight Loss (%TBWL) 6 months After Balloon Removal | 6 months
  Percentage of total body weight loss (%TBWL) will be calculated as 6 months after removal of balloon.
Change in liver enzymes | 6 months
  Liver enzymes are non-invasive markers of liver injury. Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) change will be studied in comparison with baseline levels
Number of Subjects with >= 25% Excess Body Weight Loss at 6 Months | 6 months
  Total number of patients achieving more than 25% Excess weight loss at 6 months will be studied.
Changes in Glycemic control | 6 months
  Changes in glycemic control will be assessed by change in HbA1c after 6 months of balloon removal will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Kalapala, DNB, Principal Investigator — Asian Institute of Gastroenterology
Locations (1):
- Asian Institute of Gastroenterology Hospital, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kalapala R, Jagtap N, Rughwani H, Asif S, Sekaran A, Sharma M, Kulkarni A, Rao PN, Tyagi A, Reddy DN. Adjustable Intragastric Balloon for Metabolic Dysfunction-associated Steatotic Liver Disease-Enhanced Weight Loss and Histological Improvement. J Clin Exp Hepatol. 2025 Nov-Dec;15(6):103152. doi: 10.1016/j.jceh.2025.103152. Epub 2025 Aug 12. PMID 40969863